CLINICAL TRIAL: NCT06156267
Title: An Exploratory Study of Neoantigen Personalized mRNA Vaccines in Combination With Adebrelimab and Sequential mFOLFIRINOX Regimen in Patients With Surgically Resected Pancreatic Adenocarcinoma
Brief Title: Study of Personalized Tumour Vaccines and a PD-L1 Blocker in Patients With Surgically Resected Pancreatic Adenocarcino
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Shanghai Regenelead Therapies Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Xian-Jun Yu, Principal Investigator, Fudan University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PANC-IIT-RGL-mRNA vaccine
Record Dates: First submitted 2023-11-08; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Part A: Dose Escalation, Part B: Dose Expansion (Experimental)
  Interventions: Drug: Adebrelimab; Drug: mRNA tumor vaccines

INTERVENTIONS:
Drug: Adebrelimab — Adebrelimab is a programmed death-ligand 1 antibody.
Drug: mRNA tumor vaccines — neoantigen personalized mRNA vaccines

SUMMARY:
This is a phase 1, open-label study to evaluate the safety and tolerability of neoantigen personalized mRNA tumour vaccine combined with Adebrelimab (a PD-L1 humanized monoclonal antibody) in patients with surgically resected pancreatic adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed the informed consent form and complied with protocols requirements.
2. Patients with radiographically resectable primary pancreatic tumors with histopathology or cytology confirmed resected ductal pancreatic adenocarcinoma (PDAC) with macroscopic complete resection (R0 and R1).
3. Pancreatic cancer surgical staging per AJCC 8th edition staging: T 1-3, N0-2, M0.
4. Tumour specimen availability.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
6. Life expectancy ≥ 6 months.
7. Surgical complications have recovered, or complications lower than Clavien-Dindo complication grade 3.
8. Adequate marrow and organ function.
9. Patients with fertility are willing to use an adequate method of contraception.

Exclusion Criteria:

1. Prior anti-PDAC therapy (e.g., chemotherapy, radiotherapy, targeted therapy, immunotherapy and therapeutic tumor vaccines) prior to initiation of study treatment.
2. Unsuitable for immunotherapy assessed by the investigator.
3. Plan to receive a live-attenuated vaccine within 28 days prior to initiation of study treatment or during the study treatment or within 90 days after the end of study treatment.
4. Have any active autoimmune disease, or have a history of autoimmune disease and have received systemic therapy in the past 2 years.
5. Active tuberculosis or a history of active tuberculosis infection within 28 days prior to initiation of study treatment.
6. Known or highly suspected history of interstitial pneumonia.
7. Allergic to research drug ingredients, or have a history of severe allergic reactions to other vaccines.
8. Prior malignancy within 5 years prior to study entry.
9. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
10. Known splenectomy history.
11. Concurrent severe infection within 28 days prior to initiation of study treatment.
12. Congenital or acquired immune deficiency.
13. Active hepatitis B (HBV-DNA≥1000IU/ml), hepatitis C (hepatitis C antibody positive, and HCV-RNA higher than the lower limit of assay).
14. Uncontrolled or severe cardiovascular disease.
15. Other situations that are not suitable for inclusion in this study judged by investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
DLT | Day 1 to Day 28 after the first tumour vaccine was administrated
  Percentage of subjects who meet the criteria of DLT in DLT observation period
MTD/MAD | From first dose up to end of the study, assessed up to 36 months
  Maximum tolerated dose (MTD)/Maximum administrated dose (MAD)
RDE | From first dose up to end of the study, assessed up to 36 months
  Recommended dose of expansion
AE | From date of ICF up to end of the study, assessed up to 36 months
  Percentage of subjects with Adverse Events (AEs)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pancreatic Surgery, Fudan University Shanghai Cancer Center; Pancreatic Cancer Institute, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No